CLINICAL TRIAL: NCT05789225
Title: Evaluation of a Self-management Program to Prevent Falls in Ambulatory and Non-ambulatory People With Multiple Sclerosis
Brief Title: Evaluation of a Self-management Program to Prevent Falls in People With Multiple Sclerosis
Acronym: Fewer Falls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Charlotte Ytterberg, Lecturer, associate professor (docent), Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-02553
Record Dates: First submitted 2023-03-04; First posted 2023-03-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Self-management; Accidental Falls; Health Economics; Randomized Controlled Trial; Complex Intervention; Process Evaluation; Group-based; Online Intervention; Short Message Service
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Participants will be stratified for ambulation level (ambulatory/non-ambulatory) and a 1:1 allocation ratio of blocks of 8 will be used for randomization.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fall prevention program + brochure (Experimental): Fall prevention program and brochure about falls and fall risk factors
  Interventions: Behavioral: Fall prevention program
- Brochure (Active Comparator): Brochure about falls and fall risk factors
  Interventions: Other: Brochure

INTERVENTIONS:
Behavioral: Fall prevention program — The intervention consists of the fall prevention program for ambulatory and non-ambulatory people with multiple sclerosis. The program is group-based with 8 participants in each group, led by a facilitator, and performed online. It comprises seven two-hour sessions held once a week, and a booster session held four weeks after the seventh session. In addition participants will receive a brochure about falls and fall risk factors.
  Arms: Fall prevention program + brochure
Other: Brochure — Control-group participants will receive a brochure about fall risk factors and fall prevention in addition to the standard MS care and rehabilitation.
  Arms: Brochure

SUMMARY:
The goal of this randomized controlled trial is to evaluate the effects of a digital group based self-management fall prevention program, "Fewer Falls in MS", in people with multiple sclerosis (PwMS). The main questions it aims to answer are:.

* Is the Fewer falls in MS program effective in reducing fall incidence in PwMS at 6 and 12 months after start of intervention?
* Does the program have an effect on secondary outcomes at 3, 6 and 12 months?
* How do process evaluation components (context, implementation, mechanisms of impact) inform interpretation of outcomes?
* What is the cost effectiveness of the fall prevention program 12 months after start of intervention?

Participants in the intervention group will participate in a group-based self-management fall prevention intervention of eight 2-hour sessions delivered online by a group leader. The group leader will participate in an online education program before intervention start. Home assignments are completed by the participants between group sessions. Participants in the intervention group and the control group will receive a brochure on fall risk factors and fall prevention

Researchers will compare the intervention group and the control group to see if there are any differences in fall incidence, sense of control of falls prevention, fear of falling, falls self-efficacy, activity curtailment, perceived impact of MS, self-reported health, and health economic costs. Researchers will also study factors and mechanisms that support or hinder how the fall prevention program builds participants' ability to manage their fall risk; and if and how PwMS have implemented and use self-management fall prevention behaviours into their daily lives.

DETAILED DESCRIPTION:
Purpose and aims The overall purpose is to evaluate an online fall prevention programme for ambulatory and non-ambulatory people with multiple sclerosis (PwMS). The programme incorporates key features of self-management and addresses a variety of fall risk factors. The effects of the programme in decreasing number of falls will be evaluated in a full scale randomised controlled trial (RCT). The hypothesis is that after participating in the programme, PwMS will identify and self-manage risk factors for falls in their everyday life while taking the daily fluctuations of multiple sclerosis (MS) into consideration (i.e., develop fall prevention behaviours), and thereby reduce the number of falls.

Aims:

1. To determine if the fall prevention programme is effective in reducing falls in PwMS 6 and 12 months after start of intervention.
2. To determine if the program has an effect on secondary outcomes at 3, 6 and 12 months.
3. To explore how process evaluation components (context, implementation, mechanisms of impact) inform interpretation of outcomes.
4. To evaluate the cost effectiveness of the fall prevention program at 12 months after start of intervention.

INTRODUCTION MS is a chronic inflammatory, demyelinating, and neurodegenerative disease with a global prevalence of about 36 per 100,000 population. The prevalence in women is two to four times higher than in men and the usual onset is between 20 and 40 years of age. The disease is typically progressive in nature with consequences that include an increased risk for falls. Up to 71% of PwMS fall each six months (1). Those who report a fall in the past year have an 82% probability of falling again in the six months after a fall and a 56% probability of sustaining an injurious fall (1). Falls among PwMS are associated with injuries, fear of falling and low health-related quality of life (2).

Several consequences of MS are known fall risk factors for this population, including impaired balance, reduced walking speed, and impaired cognition (2). The lack of attention given to behavioural and environmental influences on fall risk for PwMS is a major gap in existing evidence. Another major gap in MS falls research is that few studies have explored influences on fall risk among individuals who are non-ambulatory, i.e., only capable of walking a few steps or not at all (3). Furthermore, most interventions aiming to prevent falls among PwMS have excluded non-ambulatory individuals. To date, only two research teams are addressing the fall prevention needs of non-ambulatory PwMS: ours and a team based in the U.S. (4). The importance of targeting a variety of modifiable risk factors through fall prevention programs for PwMS has been highlighted (5). The need for comprehensive approaches to fall prevention that address physical, environmental, and behavioural aspects of falls management has been echoed by Gunn et al (6). Despite the recognition of the value of attention to diverse influences on fall risk, most fall prevention interventions for PwMS focus only on addressing physical impairments, such as compromised balance.

For PwMS, who live with an unpredictable disease and daily fluctuations in functioning, the benefits of self-management (7) of the multifactorial fall risks have been highlighted (8). Nevertheless, research on self-management interventions to prevent falls in PwMS is in its infancy. The delivery and settings of previous interventions have been face-to-face in physical locations, supported by online resources, or web-based without any in real-time interactions. Our proposed self-management intervention will be enhanced by digital health technologies with real-time digital meetings and online learning platforms. For PwMS, such delivery will require less time and no expenses for travelling, reduced impact on fatigue, and have the possibility to reach people also in sparsely populated areas.

The intervention To address the unique fall prevention needs of ambulatory and non-ambulatory PwMS, we have designed an online self-management fall prevention intervention. The intervention is a complex intervention, given its number of interacting components; the number and difficulty of behaviours required by both those delivering and receiving the interventions; and the number of outcomes addressed. The intervention was developed informed by findings from our scoping review (manuscript submitted), social cognitive theory (SCT) (9), and using a co-design method (10), based on design thinking (11), with the goal of enhancing the intervention's quality and relevance to end users. The co-design process (including pre-planning, the workshops, and the refinement phase) captured feedback from various stakeholders (PwMS, the patient organisation Neuro Sweden and healthcare professionals); and resulted in a manualized, online fall prevention programme.

The programme is group-based with maximum 8 participants; led by a trained facilitator; and performed in eight two-hour sessions, the first seven over seven consecutive weeks and the last final session held one month after the seventh session. The sessions are face-to-face digital meetings by use of a video platform (Zoom Video Communications, Inc.). An online learning platform (BASS) is used to share intervention content including assignments to be completed by participants between sessions, and for asynchronous activities and communication with the facilitator that can be shared between participants outside the sessions. The assignments are designed to provide participants with opportunities to practice skills learned during the fall prevention programme. One facilitator will lead each programme cycle, i.e., the eight sessions. The intervention focuses on six core self-management skills (7): problem solving, decision-making, using resources, partnership with healthcare providers, taking action, and self-tailoring. The components of the intervention are theoretically grounded in SCT (9) including observational learning, persuasion and support, and opportunities for skill mastery. The pedagogical format is theoretically grounded in universal design for learning (12) and principles for collaborative learning with blended methods (digital tools and learning platform involved) (13). Universal design for learning emphasizes the importance of designing an intervention to enable participants of various abilities to assimilate the knowledge using different forms of engagement, materials, action, and expression. The blended learning design adds to this by structuring the sessions according to principles for group collaboration in an online setting. Each of those features are reflected in the intervention.

To support program fidelity the group leaders will complete a train-the-trainer program prior to the intervention start. This online education program consists of asynchronous online modules providing information on: the fall prevention programme aim, structure, and content; theoretical grounding of the fall prevention programme; the role of the group leader; basic knowledge on MS, and on falls in MS; how to use an action plan; and detailed content of the eight session manuals. Each train-the-trainer module ends with a quiz or a reflective question. One module of the train-the-trainer program consists of a synchronous online role-play session. In addition, the group leaders will receive a manual that describes how the program's digital tools are used.

The intervention is currently evaluated in a feasibility study (14) comprising 46 participants: 23 have been randomized to participate in the group-based self-management intervention and 23 have been randomized to the control group. Analyses of feasibility of delivery of the intervention, intervention fidelity, feasibility of outcome measures, and acceptability of the intervention from the perspectives of both the PwMS who participated in the intervention and facilitators are ongoing. Preliminary findings show that the recruitment process, the data collection procedures, and the intervention procedures are feasible.

Methods Consistent with the Medical Research Council's recommendations for development and evaluation of complex interventions, the fall prevention programme will be evaluated regarding outcome and process with quantitative and qualitative methods. To ensure patient benefit, MS-specific representatives from the patient organisation Neuro Sweden have been project partners in the programme development and feasibility testing. They will continue to be project partners in this effectiveness study through ongoing collaborative discussions on project procedures, for example development of interview questions.

Effect study Aims: To determine if the fall prevention programme is effective in reducing falls in PwMS 6 months and 12 months after start of intervention; and To determine if the program has an effect on secondary outcomes at 3, 6 and 12 months.

Participants: Eligible participants will be community dwelling PwMS aged ≥ 18 years, who are able to independently transfer from bed to wheelchair with or without aids but without assistance of another person, have experienced one or more falls during the last year, are able to understand and communicate in Swedish; and have ability to use and access to cell phone and technical devices for online meetings i.e., computers or tablets with internet access. Participants will be recruited from in- and outpatient MS- and rehabilitation clinics, by the patient organization Neuro Sweden and by social media advertisements.

Power calculation: The literature suggests that 71% of PwMS fall each 6 months (1). Based on the estimation that the intervention will reduce the falls incidence to 50% in the intervention group, and allowing for approximately 15% dropout, the recruitment target is set to 104 participants in each group (80% power, p=0.05, 2-sided).

Design and procedures: A parallel-group RCT will be conducted. After informed consent, digitally collected through BASS electronic data capture tools hosted at Karolinska Institutet, participants will be allocated to intervention or control group. Participants (n=208) will be stratified for ambulation level (ambulatory/non-ambulatory) and a 1:1 allocation ratio of blocks of eight will be used. Intervention-group participants will participate in the fall prevention programme. Control-group participants will receive a brochure about fall risk factors and fall prevention in addition to the standard MS care and rehabilitation. Baseline data and follow-up assessments will be collected and managed using BASS, except short version of Montreal Cognitive Assessment which will be collected through telephone (see below). .

Approximately eight facilitators will be recruited to lead one or more cycles of the fall prevention programme in parallel groups. This will ensure that the outcomes of the programme are not attributed to an individual facilitator. The facilitators will not be involved in the usual care of the participants.

In both groups, falls will be monitored from baseline via an online short message service (SMS). An SMS will be sent once a week (to avoid recall bias) asking "Have you fallen within the last week?" Participants answering "yes" will receive a questionnaire through BASS with questions on fall related injuries. Fall is defined as "an unexpected event in which the participants come to rest on the ground, floor, or lower level". In line with recommendations for evaluation of fall prevention interventions the monitoring of falls will continue until 12 months after start of intervention.

Data-collection: Baseline data include sociodemographic (e.g., age, sex, civil status, work status) and disease-related characteristics (e.g., MS severity); expectations on the programme; self-reported falls in the previous 6 months, health literacy (HLS-EU Q16), depression/anxiety (Hospital Anxiety and Depression Scale), fatigue (Fatigue Severity Scale), cognition (short version of Montreal Cognitive Assessment), and the outcomes. Primary outcome is fall incidence. Secondary outcomes include data on self-management fall prevention behaviours assessed by the Falls Control Scale; a direct measure of fear of falling; falls self-efficacy assessed by the Revised Short Falls Efficacy Scale International, Short Falls Efficacy Scale-International (ambulatory participants) and the Spinal Cord Injury Fall Concern Scale (non-ambulatory participants); ; a direct measure of activity curtailment; perceived impact of MS assessed by the Multiple Sclerosis Impact Scale; and health status by the EuroQol-5D-5L. Data will be collected at baseline, directly after the last session, and 6 and 12 months after start of intervention.

Analyses: Intention-to-treat and per protocol analyses will be performed. Per protocol analyses will include participants who fulfil content adherence, i.e., completion of at least two action plans. Descriptive statistics will be used to present data. Linear mixed models analyses will be used for the primary outcome and normally distributed secondary outcomes. Non-parametric methods will be used for between- and within-group analyses for categorical and non-normally distributed secondary outcomes. Primary endpoint is 6 months after start of intervention. In addition, analyses of sustainability will be performed after 12 months. Analyses will be performed and reported in accordance with the Consolidated Standards of Reporting Trials guidelines for RCT. A data management plan is established and stored at the Research Data Office at Karolinska Institutet.

Process evaluation Aim: To explore how process evaluation components (context, implementation, mechanisms of impact) inform interpretation of outcomes.

Design: A mixed methods process evaluation. Participants: a) A purposively selected sample of intervention-group participants (n=20-30) to represent variation in e.g., age, sex, ambulation level, MS severity, and expectations on the programme. b) All facilitators.

Data collection: a) Semi-structured individual interviews with participants will be conducted 2- weeks, and 6- and 12-months after the end of intervention. The interviews will cover experiences of participating in the study, contextual factors and mechanisms of impact. Data from the program platform will be collected on intervention participant online activities, e.g., the action plans. b) Background information (e.g. sex, age, profession, work-related knowledge and experience). Structured questions collected after train-the-trainer and after each session covering perceived preparedness and confidence in facilitating the group, fidelity to program manual, interactions with group members, technical issues. Semi-structured interviews conducted after train-the-trainer and after the last session covering the facilitators perspective on experiences of participation, contextual factors, implementation, and mechanisms of impact.

The interviews will be conducted face-to-face or through Zoom. Analysis: Qualitative content analysis (15)- and descriptive statitics.

Health economic evaluation Aim: To evaluate the cost effectiveness of the fall prevention program at 12 months.

Participants: All intervention and control participants. Data collection: Participants answering "yes" on the weekly SMS about falls will receive a short questionnaire through BASS with questions related to fall related injuries i.e., healthcare utilization, municipal care utilization, sickness absence, medications, support from significant others, and technical aids including walking aids. Estimations of resources needed for the fall prevention program will be collected related to group facilitators i.e., time for participating in preparatory training, for conducting the program, and time for preparation in between group sessions. To estimate the monetary value of resource use, both for participants in the RCT as well as for resources needed to conduct the intervention, cost data will be retrieved from the cost per patient (KPP) database held at the Swedish Association of local authorities and regions (SKR), regional pricelists as well as from Statistics Sweden (SCB). Data on health-related quality of life will be measured using the EQ-5D-5L at all time-points.

Analyses: The PwMS participating in the new fall prevention program will be compared to the control group using intention-to-treat analysis. Descriptive and comparative statistics will be used for analyses of between and within group differences in health-related quality of life and resource use of participants as well resources needed for conducting the intervention.

Significance In contrast to previous studies of fall prevention interventions, the present is based both on pedagogical theories and on theories on behavior change; is directed to both ambulatory and non-ambulatory PwMS; and includes an interactive online design that facilitates participation from people with fatigue and those in rural areas. Thereto, most previous programmes are focused on physical activity, whereas this programme takes the multifactorial risk factors of MS falls into consideration. Through this, participants will learn strategies that they can apply in their everyday life in different fall risk areas and alter strategies as the MS progresses.

If the programme is effective in reducing the number of falls, it will be of great clinical relevance to health care providers working with PwMS. This, as well as the use of co-design in the development and use of a manualized intervention to support programme fidelity will facilitate implementation into existing health care for PwMS. We have MS-specific representatives from the patient organisation Neuro Sweden as partners which ensures the patient benefit and facilitates the dissemination of the new knowledge nationally. If effective, we will make the programme publicly available so that it can be implemented in the Swedish MS care. The generated new knowledge can also be used in Swedish national clinical guidelines for treatment of PwMS.

Key references

1. Cameron MH, Thielman E, Mazumder R, Bourdette D. Predicting falls in people with multiple sclerosis: fall history is as accurate as more complex measures. Mult Scler Int. 2013;2013:496325.
2. Coote S, Comber L, Quinn G, Santoyo-Medina C, Kalron A, Gunn H. Falls in People with Multiple Sclerosis: Risk Identification, Intervention, and Future Directions. Int J MS Care. 2020;22(6):247-55.
3. Ytterberg C, Einarsson U, Holmqvist LW, Peterson EW. A population-based study of fall risk factors among people with multiple sclerosis in Stockholm county. J Rehabil Med. 2013;45(5):452-7.
4. Rice LA, Isaacs Z, Ousley C, Sosnoff J. Investigation of the Feasibility of an Intervention to Manage Fall Risk in Wheeled Mobility Device Users with Multiple Sclerosis. Int J MS Care. 2018;20(3):121-8.
5. Sosnoff JJ, Sung J. Reducing falls and improving mobility in multiple sclerosis. Expert Rev Neurother. 2015;15(6):655-66.
6. Gunn H, Andrade J, Paul L, Miller L, Creanor S, Stevens K, et al. A self-management programme to reduce falls and improve safe mobility in people with secondary progressive MS: the BRiMS feasibility RCT. Health Technol Assess. 2019;23(27):1-166.
7. Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003;26(1):1-7.
8. Gunn H, Cameron M, Hoang P, Lord S, Shaw S, Freeman J. Relationship Between Physiological and Perceived Fall Risk in People With Multiple Sclerosis: Implications for Assessment and Management. Arch Phys Med Rehabil. 2018;99(10):2022-9.
9. Bandura A. Social foundations of thought and action: A social cognitive theory. Englewood Cliffs, New Jersey: Prentice-Hall; 1986.
10. Bate P, Robert G. Experience-based design: from redesigning the system around the patient to co-designing services with the patient. Qual Saf Health Care. 2006;15(5):307-10.
11. Carlgren L, Rauth I, Elmquist M. Framing Design Thinking: The Concept in Idea and Enactment. Creat Innov Manag. 2016;25(1):38-57.
12. Meyer A, Rose DH, Gordin D. Universal design for learning: Theory and practice. Wakefield, USA: CAST Professional Publishing; 2014.
13. Hrastinski S. What Do We Mean by Blended Learning? TechTrends. 2019;63(5):564-9.
14. Kierkegaard M, Peterson E, Tuvemo Johnson S, Gottberg K, Johansson S, Elf M, et al. Online self-management fall prevention intervention for people with multiple sclerosis: a feasibility study protocol of a parallel group randomised trial. BMJ open. 2022;12(7):e061325.
15. Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004;24(2):105-12.

ELIGIBILITY:
Inclusion Criteria:

* PwMS aged ≥ 18 years
* Able to walk or independently transfer from bed to chair or wheelchair with or without aids but without assistance of another person
* Have experienced one or more falls during the last year
* Able to understand and communicate in Swedish
* Self-rated ability to use and access to technical devices for online meetings i.e., computers or tablets with internet access and mobile phones to receive and send short message service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Falls incidence | 6 and 12-months after start of intervention
  Falls will be monitored weekly via an online short message service. A lower number of falls means a better outcome

SECONDARY OUTCOMES:
Falls Control Scale | 3, 6 and 12-months after start of intervention
  Questionnaire that includes four statements with which the participants agree or disagree on a scale from 1 to 4 where a higher score indicates better falls control.
Measure of fear of falling | 3, 6 and 12-months after start of intervention
  Questionnaire with one question "Are you afraid of falling?" and five response options: Not at all afraid, Somewhat afraid, Fairly afraid, Very afraid, Extremely afraid
Falls Efficacy Scale-International | 3, 6 and 12-months after start of intervention
  Questionnaire that consists of 16 questions regarding 'how concerned' the person is when performing daily activities. Each question is answered with a four-graded scale (1-4); not at all concerned, somewhat concerned, fairly concerned and very concerned. A total score is calculated and ranges from 16 to 64, higher scores indicate worse outcome.
Spinal Cord Injury Fall Concern Scale | 3, 6 and 12-months after start of intervention
  Questionnaire that addresses concern about falling during 16 activities of daily living associated with falling, scored on a 4-point scale (1=not at all concerned to 4=very concerned. The total score is calculated by summing the scores for each activity, with a possible range between 16 and 64, higher scores indicate worse outcome.
Revised version of the Short Falls Efficacy Scale-International | 3, 6 and 12-months after start of intervention
  Questionnaire that consists of seven questions regarding 'how concerned' the person is when performing daily activities. Each question is answered with a four-graded scale (1-4); not at all concerned, somewhat concerned, fairly concerned and very concerned. A total score is calculated and ranges from 7 to 27, higher scores indicate worse outcome.
Activity curtailment | 3, 6 and 12-months after start of intervention
  Questionnaire with one question "Do you think fear of falling has made you cut down on any activities that you used to do?" with four response options: Yes, No, Don't know, Refuse to answer
Multiple Sclerosis Impact Scale | 3, 6 and 12-months after start of intervention
  Questionnaire - 29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of multiple sclerosis on day-to-day life in the past two weeks. All items have 5 response options: 1 "not at all" to 5"extremely". Each of the two scales are scored by summing the responses across items, then converting to a 0-100 scale where 100 indicates greater impact of disease, i.e. worse outcome.
EuroQol-5D-5L | 3, 6 and 12-months after start of intervention
  Questionnaire consisting of the EQ-5D Index and the EQ Visual Analogue Scale. The EuroQol 5D-5L comprises five pre-defined dimensions: Mobility, Self-care, Usual activities, Pain/discomfort and Anxiety/depression. The respondent rates each dimension on a five level scale as having no problem, slight problems, moderate problem, severe problem, unable or extreme. The answers are then converted to an index value (the EQ Index) ranging from 0 (representing death) to 1 (full health). The EQ VAS records the respondent's self-rated health on a 20-centimeter vertical visual analo,g scale with end-points ranging from 0 to 100. The single global question in the EQ VAS asks the individual to label his/her health as "the worst health you can imagine" (0) to "the best health you can imagine"

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Ytterberg, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results in a publication, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately following publication and ending two years after publication
Access Criteria: Since data can indirectly be traced back to the study participants, according to the Swedish and EU personal data sharing legislation, access can only be granted upon request. Request for access to the data can be put to our Research Data Office (rdo@ki.se) at Karolinska Institutet, and will be handled according to the relevant legislation. In most cases, this will require a data processing agreement or similar with the recipient of the data.

REFERENCES:
- [Background] Tuvemo Johnson S, Flink M, Peterson E, Gottberg K, Elf M, Johansson S, Kierkegaard M, Ytterberg C. Self-management of falls in people with multiple sclerosis: A scoping review. Clin Rehabil. 2023 Feb;37(2):162-176. doi: 10.1177/02692155221128723. Epub 2022 Sep 29. PMID 36177511
- [Background] Kierkegaard M, Peterson E, Tuvemo Johnson S, Gottberg K, Johansson S, Elf M, Flink M, Ytterberg C. Online self-management fall prevention intervention for people with multiple sclerosis: a feasibility study protocol of a parallel group randomised trial. BMJ Open. 2022 Jul 8;12(7):e061325. doi: 10.1136/bmjopen-2022-061325. PMID 35803627
- [Background] Tuvemo Johnson S, Flink M, Gottberg K, Walker Peterson E, Meijer U, Bylinder J, Kierkegaard M, Ytterberg C. Effectiveness of Fewer Falls, an online group-based self-management fall prevention programme for people with multiple sclerosis: protocol of a randomised controlled trial. BMJ Open. 2025 Jan 6;15(1):e089217. doi: 10.1136/bmjopen-2024-089217. PMID 39762097
- [Background] Johnson ST, Ytterberg C, Peterson E, Johansson S, Kierkegaard M, Gottberg K, Flink M. Development of Fewer Falls in MS-An Online, Theory-Based, Fall Prevention Self-Management Programme for People With Multiple Sclerosis. Health Expect. 2024 Aug;27(4):e14154. doi: 10.1111/hex.14154. PMID 39032151
- [Background] Meijer U, Flink M, Tuvemo Johnson S, Kierkegaard M, Gottberg K, Ytterberg C. Preventing falls in multiple sclerosis: a qualitative study on user requirements for a self-management programme. Disabil Rehabil. 2025 Jan;47(2):398-405. doi: 10.1080/09638288.2024.2348725. Epub 2024 May 7. PMID 38711397